CLINICAL TRIAL: NCT06979232
Title: Enhanced White Light Endoscopy Versus Conventional White Light Endoscopy for Colorectal Adenoma Detection: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: LY2024-320-C
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Adenoma
Keywords: Enhanced white light endoscopy; Adenoma detection rate; Randomized controlled trial

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-WLI (Experimental): Enhanced White Light Imaging
  Interventions: Device: Enhanced White Light Imaging
- WLI (Placebo Comparator): White Light lmaging
  Interventions: Device: White Light lmaging

INTERVENTIONS:
Device: Enhanced White Light Imaging — Use of E-WLI for colon inspection during both insertion and withdrawal phase of colonoscopy
  Arms: E-WLI
Device: White Light lmaging — Use of WLl for colon inspection during both insertion and withdrawal phase of colonoscopy
  Arms: WLI

SUMMARY:
1. Study on Adenoma Detection Rate (ADR) Comparing Enhanced White Light Endoscopy (E-WLI) versus Conventional White Light Endoscopy (WLI);
2. Study Comparing Enhanced White Light Endoscopy (E-WLI) versus Conventional White Light Endoscopy (WLI) for Detection Rates of Sessile Serrated Lesions (SSLs), Total Polyp Detection Rate, and Advanced Adenoma Detection Rate;
3. Study on Polyp Characteristics (Size, Location, etc.) Observed Using Conventional White Light Endoscopy (WLI) and Enhanced White Light Endoscopy (E-WLI).

DETAILED DESCRIPTION:
Before colonoscopy, gastroenterology specialists stratified eligible patients according to 1) colorectal cancer screening, 2) positive fecal immunochemical test (FIT) results or gastrointestinal symptoms, and 3) follow-up colonoscopy after colorectal polyp treatment. Patients were then randomized in a 1:1 ratio to receive either colonoscopy with enhanced white light imaging (E-WLI group) or high-definition conventional white light imaging (WLI group) during both insertion and withdrawal phases. Randomization was based on random number lists generated by the coordinating center for each participating site. Endoscopists performing the procedures were not involved in generating the randomization sequence. All procedures were performed by experienced endoscopists at participating centers (>2000 colonoscopy screenings). All procedures utilized endoscopes with "Xiaohua Tanying" technology that incorporated E-WLI functionality. Bowel preparation was assessed and graded by the performing endoscopist using the Boston Bowel Preparation Scale (BBPS). Endoscopy specialists and healthcare facility staff followed standard procedures for patient management and monitoring, including anesthesia. Cecal intubation was verified by the endoscopist through photographic documentation identifying the ileocecal valve and appendiceal orifice. Insertion and withdrawal times were measured through video recording analysis, excluding time spent on therapeutic interventions and washing. Endoscopists were required to maintain a minimum withdrawal inspection time of 6 minutes (with at least 2 minutes each for right colon, transverse colon, and left colon). Regardless of group assignment (E-WLI or WLI), when polyps were detected during the procedure, they were observed using both WLI and E-WLI (2 modes), with images captured in each mode. The location, size, and morphology (Paris classification) of all polyps were documented. All polyps were removed (or biopsied if unresectable), and pathological results were obtained. For hyperplastic polyps in the rectum, if more than 3 diminutive polyps were present, only the first 3 detected polyps required management.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female aged 45 to 85
* 2. Patients undergoing colonoscopy for colorectal cancer screening, positive fecal immunochemical test (FIT) results, gastrointestinal symptoms, or follow-up examination after colorectal polyp treatment
* 3. Capable of providing informed consent and agreeing to participate
* 4. Able and willing to follow all research processes

Exclusion Criteria:

* 1. Participated in other clinical trials, signed informed consent form, and in the follow-up period of other clinical trials;
* 2. Participated in clinical trials of drugs and is in the discontinuation period of experimental or control drugs;
* 3. Have had drug or alcohol abuse or psychological disorders in the past five years.
* 4. Pregnant or lactating patients;
* 5. Known to have polyposis syndrome;
* 6. Patients with gastrointestinal bleeding;
* 7. Previous history of inflammatory bowel disease, colorectal cancer, or colorectal surgery;
* 8.Patients with contraindications to tissue biopsy;
* 9. History of allergies to the ingredients in intestinal cleansers;
* 10. Individuals with conditions such as intestinal obstruction or perforation, toxic megacolon, heart failure (grade III or IV), severe cardiovascular disease, severe liver failure, or renal insufficiency, among others.
* 11. Researchers believe that patients are not suitable to participate in the trial.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate (ADR) | 14 days
  ADR was calculated by dividing the total number of patients detected with adenomas by the total number of patients who underwent colonoscopy

SECONDARY OUTCOMES:
Polyp Detection Rate(PDR) | 14 days
  Calculated by dividing the total number of patients with detected polyps by the total number of patients undergoing colonoscopy.
Sessile serrated lesion detection rate (SDR) | 14 days
  SSLDR was calculated by dividing the total number of patients detected with sessile serrated lesions by the total number of patients who underwent colonoscopy.
Advanced Adenoma Detection Rate (aADR) | 14 days
  Calculated by dividing the total number of patients with detected advanced adenomas by the total number of patients undergoing colonoscopy.
Mean number of polyps per patient (MPP) | 14 days
  Calculated by dividing the total number of detected polyps by the total number of patients undergoing colonoscopy.
Mean number of Adenomas per patient(MAP) | 14 days
  Calculated by dividing the total number of detected adenomas by the total number of patients undergoing colonoscopy.
Detection Rate of Polyps of Different Sizes | 14 days
  lt is calculated by dividing the number of patients with polyps with different sizes by the total number of patients undergoing colonoscopy.
Detection Rate of Adenomas with Different Morphologies | 14 days
  lt is calculated by dividing the number of patients with adenomas of different morphologies by the total number of patients undergoing colonoscopy.
Average Number of Adenomas with Different Morphologies | 14 days
  lt is calculated by dividing the number of adenomas with different morphologies by the total number of patients undergoing colonoscopy.
Average Number of Polyps of Different Sizes | 14 days
  lt is calculated by dividing the number of polyps with different sizes by the total number of patients undergoing colonoscopy.
Detection Rate of Adenomas of Different Sizes | 14 days
  lt is calculated by dividing the number of adenomas with different sizes by the total number of patients undergoing colonoscopy.
Average Number of Adenomas of Different Sizes | 14 days
  lt is calculated by dividing the number of adenomas with different sizes by the total number of patients undergoing colonoscopy.
Detection Rate of Adenomas in Different Locations | 14 days
  lt is calculated by dividing the number of patients with detected adenomas in different locations by the total number of patients undergoing colonoscopy.
Average Number of Adenomas in Different Locations | 14 days
  lt is calculated by dividing the number of detected adenomas in different locations by the total number of patients undergoing colonoscopy.
Detection Rate of Polyps in Different Locations | 14 days
  lt is calculated by dividing the number of patients with polyps in different locations by the total number of patients undergoing colonoscopy.
Average Number of Polyps in Different Locations | 14 days
  lt is calculated by dividing the number of detected polyps in different locations by the total number of patients undergoing colonoscopy.
Detection Rate of Polyps with Different Morphologies | 14 days
  lt is calculated by dividing the number of patients with polyps of different morphologies by the total number of patients undergoing colonoscopy.
Average Number of Polyps with Different Morphologies | 14 days
  lt is calculated by dividing the number of polyps with different morphologies by the total number of patients undergoing colonoscopy.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - The First People's Hospital of Lanzhou City, Lanzhou, Gansu
  - The Third Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Armed Police Forces Hospital of Sichuan, Leshan, Sichuan
  - People's Hospital of Bayingolin Mongol Autonomous Prefecture, Korla, Xinjiang
  - Ningbo Ninth Hospital, Ningbo, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No